CLINICAL TRIAL: NCT01936649
Title: A Phase 4, Open-label Test-retest Study to Assess the Reproducibility of Quantitative Measurements of Myocardial Uptake of AdreView (Iobenguane I 123 Injection)
Brief Title: Open-label, Test-retest Study Assessing Reproducibility of Quantitative Measurements of Myocardial Uptake of AdreView.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GE Healthcare (Industry)
Collaborators: H2O Clinical LLC (Industry); Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GE-122-015
Record Dates: First submitted 2013-09-03; First posted 2013-09-06 (Estimated); Results first posted 2015-01-26 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-10

CONDITIONS: Heart Failure (HF); Ventricular Dysfunction, Left
Keywords: Nuclear imaging; Radiopharmaceutical; Iobenguane; I-123; reproducibility; Quantitative measurements; myocardial uptake; SPECT imaging; planar imaging; AdreView™
MeSH Terms: conditions — Heart Failure; Ventricular Dysfunction, Left | interventions — 3-Iodobenzylguanidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AdreView (Iobenguane I 123 Injection) (Experimental): Two administrations of single intravenous (i.v) injection of Iobenguane I 123 10 millicuries (mCi) (370 MBq) over 1 to 2 minutes within an interval of 5 to 14 days.
  Interventions: Drug: AdreView (Iobenguane I 123 Injection)

INTERVENTIONS:
Drug: AdreView (Iobenguane I 123 Injection) — AdreView 10 mCi as a single i.v administration
  Other Names: meta-iodobenzylguanidine (123 I-mIBG)

SUMMARY:
The aim of the study was to assess the reproducibility of quantitative measurements of myocardial uptake of Iobenguane I 123 on planar and single photon emission computed tomography (SPECT) imaging following intravenous (i.v.) administration of AdreView. Efficacy was assessed based upon the absolute differences between quantitative analyses of imaging data on 2 scans performed 5 to 14 days apart.

ELIGIBILITY:
Inclusion Criteria:

* The participant was originally diagnosed with New York Heart Association (NYHA) Class II-III HF due to ischemic heart disease at least 3 months or due to non-ischemic cardiomyopathy at least 6 months before enrollment into the study.
* The participant had Left Ventricular (LV) dysfunction with Left Ventricular Ejection Fraction (LVEF) less than or equal to 35% measured by an appropriate method (e.g., radionuclide or contrast ventriculography, electrocardiogram [ECG]-gated SPECT myocardial perfusion imaging [MPI], magnetic resonance [MR] imaging, computed tomography [CT] or echocardiography) within 6 months of enrollment into the study and documented in the participant's medical record.
* The participant had a history of compliance with prescribed heart failure (HF) medications and took HF guidelines-based medication at study entry including at a minimum a beta-blocker and either an angiotensin converting enzyme inhibitor or angiotensin receptor antagonist unless documented to be intolerant to any of these classes of medications.
* The participant had been on a stable medical regimen for a minimum of 3 months, with no hospitalizations or change in HF medications or HF symptoms.
* Participants must be clinically stable for at least 7 days before enrolling into the study (e.g., not experiencing continuing chest pain or hemodynamic instability).

Exclusion Criteria:

* The participant had previously received 123 I-mIBG or 131 I-mIBG.
* The participant had known or suspected hypersensitivity/allergy to iodine, Iobenguane or to any of the excipients in AdreView.
* The participant had a heart transplant at any time prior to enrollment.
* The participant had LVEF >35% as measured by an appropriate method (e.g., radionuclide or contrast ventriculography, ECG-gated SPECT MPI, MR, CT, or echocardiography) within 30 days prior to enrollment into the study.
* The participant had received defibrillation either external or via an implantable cardioverter defibrillator (ICD), anti-tachycardia pacing, or cardioversion to treat an arrhythmic event in the previous 90 days.
* The participant had a cardiac revascularization, insertion of an ICD, or acute myocardial infarction within 30 days before study entry.
* The participant used any of the following medications: Amitriptyline and derivatives, imipramine and derivatives, other antidepressants that inhibit the norepinephrine transporter, antihypertensives that deplete norepinephrine stores or inhibit reuptake, sympathomimetic amines and cocaine.
* The participant had either NYHA Class I or NYHA Class IV HF at the time of study entry.
* The participant had renal insufficiency (creatinine >3 mg/dl).
* The participant had participated in a clinical trial involving IMP or devices within 30 days prior to first administration of AdreView™.
* In the investigator's opinion, the participant's medical history included either extensive lifetime exposure to ionizing radiation (medical, occupational, other) or documented total radiation dose >50 mSv during the previous 5 years.
* The participant had experienced HF hospitalization, increased HF symptoms without hospitalization, or had a change or increase in HF medications during the previous 3 months.
* The participant had a serious non-cardiac medical condition associated with significant elevation of plasma catecholamines, including pheochromocytoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2013-08; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arnold Jacobson, M.D., Study Chair — GE Healthcare
Locations (1):
- GE Healthcare, Princeton, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 10 centers in US. A total of 63 participants were enrolled in the study between 16 August 2013 and 20 February 2014.
Pre-assignment Details: Out of 63 enrolled participants, 51 received at least 1 administration of AdreView (Iobenguane I 123 injection) and 50 participants received 2 administrations of AdreView. Myocardial AdreView uptake over time was quantitatively measured via planar and single photon emission computed tomography (SPECT) imaging at various time points post-injection.
Groups:
- AdreView (Iobenguane I 123 Injection): Two administrations of single intravenous (i.v.) injection of Iobenguane I 123 10 millicuries (mCi) (370 MBq) over 1 to 2 minutes within an interval of 5 to 14 days.
Period: Overall Study
Arm/Group | AdreView (Iobenguane I 123 Injection)
Started | 63
Treated | 51
Completed | 50
Not Completed | 13
Not completed — Withdrawal by Subject | 4
Not completed — Physician Decision | 2
Not completed — Protocol Violation | 2
Not completed — Other than specified above | 5

BASELINE CHARACTERISTICS:
Population: Safety population defined as all enrolled participants who received at least 1 administration of AdreView (Iobenguane I 123 Injection).
Groups:
- AdreView (Iobenguane I 123 Injection): Two administrations of single i.v. injection of Iobenguane I 123 10 mCi (370 MBq) over 1 to 2 minutes within an interval of 5 to 14 days.
Arm/Group | AdreView (Iobenguane I 123 Injection)
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (12.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 43
Region of Enrollment [Number; unit: participants]
  United States | 51
Safety Assessment [Number; unit: participants] | 51

OUTCOME MEASURES:

1. Primary Outcome: To Assess Test-retest Reproducibility of Iobenguane I 123 Injection Myocardial Uptake in Heart Failure (HF) Participants on Planar Imaging at 3 Hours 50 Minutes Following I.V. Injection of AdreView (Iobenguane I 123 Injection)
Description: Participants underwent 2 AdreView (Iobenguane I 123 Injection) exams on the same gamma camera within 5 to 14 days, with the requirement that there was no change in the clinical condition of the participant or in the imaging equipment between the 2 procedures. Each imaging study was processed and read independently by 3 technologists. Mean heart/mediastinum (H/M) ratio difference (with 95% confidence interval [CI]) was used as the measure of test stability.
Time Frame: 3 Hours 50 Minutes post administration of 2 dosing within an interval of 5 to 14 days
Population: Efficacy population that included all participants who underwent 2 administrations of AdreView (Iobenguane I 123 Injection); had at least an interpretable planar image acquisition at 3 hours 50 minutes post-injection after each AdreView administration. Here, 'n' signifies number of participants analyzed by the technologist.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | AdreView (Iobenguane I 123 Injection)
Number analyzed (Participants) | 47
Ratio
  Technologist A (post dosing-1) (n=46) | 1.435 (0.2238)
  Technologist A (post dosing-2) (n=47) | 1.422 (0.2229)
  Technologist A(Dosings:absolute difference) (n=46) | 0.070 (0.0612)
  Technologist B (post dosing-1) (n=47) | 1.430 (0.220)
  Technologist B (post dosing-2) (n=47) | 1.436 (0.2069)
  Technologist B(Dosings:absolute difference) (n=47) | 0.060 (0.0413)
  Technologist C (post dosing-1) (n=47) | 1.427 (0.2115)
  Technologist C (post dosing-2) (n=47) | 1.441 (0.1945)
  Technologist C(Dosings:absolute difference) (n=47) | 0.067 (0.0537)
  Average (post dosing-1) (n=47) | 1.429 (0.2160)
  Average (post dosing-2) (n=47) | 1.433 (0.2048)
  Average (Dosings:absolute difference) (n=47) | 0.065 (0.0348)

2. Secondary Outcome: To Assess the Test-retest Reproducibility of Iobenguane I 123 Injection Myocardial Uptake on Planar Imaging at 15 Minutes Following Administration of AdreView (Iobenguane I 123 Injection)
Description: Measurements of H/M ratio and the extent of difference between H/M measurements following AdreView administration and 15 minutes delayed planar imaging on 2 separate days within an interval of 5 to 14 days, was used to assess the test-retest reproducibility. Data from test-retest study was used to estimate the normal ranges for variation in quantitation of myocardial tracer uptake using AdreView. H/M ratios were calculated by 3 technologists and average of 3 technologists was calculated based on non-missing technologists reviewing results. All non-missing technologist evaluations were averaged per participant.
Time Frame: 15 minutes post administration of 2 dosing within an interval of 5 to 14 days
Population: Efficacy population that included all participants who underwent 2 administrations of AdreView; had at least an interpretable planar image acquisition at 15 minutes post-injection after each AdreView administration. Here, 'n' signifies number of participants analyzed by the technologist.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | AdreView (Iobenguane I 123 Injection)
Number analyzed (Participants) | 47
Ratio
  Technologist A (post dosing-1) (n=47) | 1.584 (0.2258)
  Technologist A (post dosing-2) (n=47) | 1.567 (0.2267)
  Technologist A(Dosings:absolute difference) (n=47) | 0.081 (0.0765)
  Technologist B (post dosing-1) (n=47) | 1.568 (0.2262)
  Technologist B (post dosing-2) (n=47) | 1.553 (0.2169)
  Technologist B(Dosings:absolute difference) (n=47) | 0.062 (0.0532)
  Technologist C (post dosing-1) (n=47) | 1.593 (0.2227)
  Technologist C (post dosing-2) (n=47) | 1.571 (0.2203)
  Technologist C(Dosing:absolute difference) (n=47) | 0.071 (0.0541)
  Average (post dosing-1) (n=47) | 1.581 (0.2212)
  Average (post dosing-2) (n=47) | 1.564 (0.2195)
  Average (Dosings:absolute difference) (n=47) | 0.072 (0.0485)

ADVERSE EVENTS:
Time Frame: From Baseline up to discharge from hospital on each dosing.
Description: Adverse events (AEs) reported were treatment emergent adverse events (TEAEs) that were AEs that begins (or a pre-existing AE that worsens) after receiving investigational medicinal product through the time of discharge on each dosing day.
Arm/Group | AdreView (Iobenguane I 123 Injection)
Serious Adverse Events (participants affected / at risk) | 0/51
Other Adverse Events (participants affected / at risk) | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI and/or institution is that the Sponsor can review results communications prior to public release and can restrict communications regarding trial results for a period that is more than 30 days (publications/abstracts) but not to exceed 90 days (patent related issues) from the time submitted to the Sponsor to review. The PI may be asked to remove any Sponsor confidential information and/or delay publication to protect any proprietary information.